CLINICAL TRIAL: NCT06897644
Title: Gemcitabine Plus Nab-PAclitaxel as Switch maiNTEnance Versus cONtinuation of Modified FOLFIRINOX as First-line Chemotherapy in Patients With Advanced Pancreatic Cancer: the PANThEON Phase III Trial
Brief Title: Gemcitabine Plus Nab-paclitaxel as Switch Maintenance Versus Continuation of Modified FOLFIRINOX as 1st Line Chemotherapy in Patients With Advanced Pancreatic Cancer.
Acronym: PANThEON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANThEON; 2024-515214-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma Advanced or Metastatic
Keywords: first line; mFOLFIRINOX; chemotherapy; pancreas; Gemcitabine with Nab-Paclitaxel; switch maintenance; pancreatic cancer
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A - continuation of mFOLFIRINOX (Active Comparator): Patients in Arm A will receive continuation of the same regimen used as induction chemotherapy:
  * Oxaliplatin 85 mg/sqm;
  * Irinotecan 150 mg/sqm;
  * Leucovorin 400 mg/sqm (racemic) or l-Leucovorin 200 mg/sqm;
  * 5-FU 2400 mg/sqm 46-hours infusion; every 2 weeks. Treatment will continue until PD, unacceptable toxicity, informed consent withdrawal, or patient's death.
  In case of permanent discontinuation of one or more compounds due to unacceptable toxicity, treatment with the other agent(s) may be continued until PD.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan (CPT-11); Drug: Leucovorin; Drug: 5-FU (5-fluorouracil)
- ARM B - switch maintenance with Gem-NabP (Experimental): Patients in Arm B will receive:
  * Gemcitabine 1000 mg/sqm on Days 1,8,15 of every 28-day cycles;
  * Nab-Paclitaxel 125 mg/sqm on Days 1,8,15 of every 28-day cycles. Treatment will continue until PD, unacceptable toxicity, informed consent withdrawal, or patient's death.
  In case of permanent discontinuation of one compound due to unacceptable toxicity, treatment with the other agent may be continued until PD in each arm.
  Interventions: Drug: gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Oxaliplatin — 85 mg/sqm iv over 2 hours day 1
  Arms: ARM A - continuation of mFOLFIRINOX
Drug: Irinotecan (CPT-11) — 150 mg/sqm iv over 60 minutes day 1
  Arms: ARM A - continuation of mFOLFIRINOX
Drug: Leucovorin — Leucovorin 400 mg/sqm (racemic) or l-Leucovorin 200 mg/sqm over 2 hours day 1
  Arms: ARM A - continuation of mFOLFIRINOX
Drug: 5-FU (5-fluorouracil) — 2400 mg/sqm 46-hours infusion
  Arms: ARM A - continuation of mFOLFIRINOX
Drug: gemcitabine — 1000 mg/sqm over 30 minutes on Days 1,8,15 of a 28-day cycles
  Arms: ARM B - switch maintenance with Gem-NabP
Drug: Nab-paclitaxel — 125 mg/sqm over 30 minutes on Days 1,8,15 of a 28-day cycles
  Arms: ARM B - switch maintenance with Gem-NabP

SUMMARY:
PANThEON is a randomized, open-label, multicenter phase III trial aimed at comparing the switch maintenance with gemcitabine plus nab-paclitaxel (ARM B) versus mFOLFIRINOX continuation (ARM A) in terms of overall survival (OS) in patients with unresectable LAD or mPDAC without disease progression following 3 months of induction mFOLFIRINOX triplet chemotherapy.

DETAILED DESCRIPTION:
PANThEON is a randomized, open-label, multicenter phase III trial of switch maintenance with gemcitabine plus nab-paclitaxel (ARM B) versus mFOLFIRINOX continuation (ARM A) in patients with unresectable LAD or mPDAC without disease progression following 3 months of induction mFOLFIRINOX triplet chemotherapy.

The induction chemotherapy regimen will be mFOLFIRINOX as per standard of care. Treatment must be continued for up to a maximum of 14 weeks, corresponding to ~ 6 bi-weekly cycles. A minimum of 4 treatment cycles administered is necessary for the patient to be evaluable for randomization.

Radiological tumor assessment will be performed before the start and after completion of induction chemotherapy. Patients with complete/partial response or stable disease (CR/PR/SD) or without evidence of progressive disease (PD) in case of non-measurable disease will be randomized in a 1:1 ratio.

Stratification factors will be ECOG Performance status (PS, 0 vs 1) and disease extension (LAD vs metastatic with presence of liver metastases vs metastatic without presence of liver metastases).

ELIGIBILITY:
Inclusion Criteria:

* Patient able and willing to provide written informed consent and to comply with the study protocol.
* Subjects must be ≥18 years.
* Histologically or cytologically confirmed unresectable locally advanced or metastatic pancreatic adenocarcinoma eligible for treatment in the first-line setting.
* Presence of measurable or non-measurable disease assessed by CT scan and/or MRI according to RECIST 1.1. Note: any lesion which has been subjected to percutaneous therapies or radiotherapy should not be considered measurable, unless the lesion has clearly progressed since the procedure.
* Availability of archival tumor sample (primary tumor or metastatic site) for biomarker analysis.
* ECOG performance status of 0-1 (if age < 70 years). If age ≥70 years, ECOG PS must be 0.
* Estimated life expectancy > 3 months.
* Adequate baseline hematologic function characterized by the following at screening:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L.
  * Platelets count ≥ 100 × 109/L.
  * Hemoglobin ≥ 9 g/dl. Note: prior transfusions for patients with low hemoglobin are allowed.
* Adequate liver function characterized by the following at screening:

  * Serum total bilirubin ≤ 1.5 × ULN and < 2 mg/dL. Note: Subjects with Serum total bilirubin ≥ 1.5 × ULN and conjugated bilirubin ≤ ULN or < 40% of total bilirubin are allowed.
  * Serum transaminases (AST and/or ALT) < 3 x ULN (< 5 x ULN in presence of liver metastasis). In participants with elevated AST or ALT, the values must be stable for at least 2 week and with no evidence of biliary obstruction by imaging.
* Adequate renal function, i.e. serum creatinine ≤ 1.5 x institutional ULN and calculated by Cockroft-Gault formula or directly measured creatinine clearance ≥ 50 mL/min.
* Adequate coagulation functions as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy).
* No presence of complete dihydropyrimidine dehydrogenase (DPYD) enzyme deficiency (homozygous of the following DPYD polymorphisms: c1679GG, c1905+1AA, c2846TT) with DPYD gene testing mandatory at screening as per national guidelines. UDP-glucuronosyltransferase 1A1 (UGT1A1) testing is not mandatory. However, if UGT test is routinely performed in the participating centers, enrolment of patients carriers of variants of DPYD and homozygous variant UGT1A1 [7/7] has to be discussed with the Sponsor.
* Women of childbearing potential must agree to remain abstinent (refrain from sexual intercourse) or use highly effective contraceptive methods, as defined in APPENDIX V of the full protocol, during the treatment period and for at least 7 months after the last administration of study treatments.
* Negative serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women <1 year after the onset of menopause.
* Men must agree to remain abstinent (refrain from sexual intercourse) or use highly effective contraceptive methods during the treatment period and for at least 7 months after the last administration of study treatments.
* Participants must agree not to donate eggs/sperm for future use for the purposes of assisted reproduction during the study and for a period of 7 months after receiving the last dose of study treatment. Female and male participants should consider preservation of eggs/sperm prior to study treatment as anti-cancer treatments may impair fertility.

Exclusion Criteria:

* Pancreatic neuroendocrine, acinar, squamous/adenosquamous, or islet tumors.
* Previous or concurrent systemic (e.g. cytotoxic or targeted or other experimental drugs) therapy for advanced pancreatic adenocarcinoma.

Note: previous (neo)adjuvant or perioperative anti-cancer therapy for non-metastatic, resectable or borderline resectable PDAC, associated with surgery on the primary tumor, is allowed if > 9 months have elapsed from the last dose of therapy and documented disease progression or relapse.

* Major surgery or radiation therapy performed within <4 weeks before randomization. Palliative radiotherapy to bone lesions is allowed if performed > 2 weeks prior to start of study treatment. Patients must have recovered from an effect from major surgery.
* Known allergy or hypersensitivity to study drugs and/or their excipients.
* Unresolved toxicity ≥ CTCAE grade 2 attributed to any prior therapies (e.g. grade ≥2 peripheral neurotoxicity), excluding anemia or alopecia.
* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that requires directed therapy (such as radiotherapy or surgery) or increasing doses of corticosteroids 2 weeks prior to study entry. Participants with treated symptomatic brain metastases should be neurologically stable for 4 weeks post-treatment and prior to study entry.
* Any known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years prior to study entry except for curatively treated basal cell carcinoma of the skin, in situ carcinoma of the cervix, and prostate cancer.
* Know active uncontrolled hepatitis B or hepatitis C. Patients with a past or resolved HBV infection are eligible. Patients with chronic disease controlled by antiviral therapy or requiring prophylactic treatment are eligible.
* Chronic or current active infectious disease requiring systemic antibiotics or antifungal treatment within 2 weeks prior to enrollment.
* Known uncontrolled HIV infection. HIV-positive patients are eligible if their CD4+ cell count amounts to 300 cells per μL or more; HIV viral load must be undetectable per standard of care assay, and patients must be compliant with antiretroviral treatment.
* Pregnant or breast-feeding patient, or patient planning to become pregnant within 7 months after the end of treatment.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA > II, unstable angina pectoris, history of myocardial infarction within 3 months before study entry, significant arrhythmia).
* Presence of psychiatric disorder precluding understanding of information of trial related topics and giving informed consent.
* Any serious underlying medical conditions (judged by the investigator), that could impair the ability of the patient to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | from date of randomization to date of death (or last follow up for alive patients), assessed up to 48 months
  OS is defined as the time from randomization to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | from randomization to disease progression or death from any cause, assessed up to 48 months
  PFS will be defined as the time from randomization until disease progression or death, whichever will occur first; for patients alive and without progression time will be censored at the last known follow-up.
Time to Treatment Failure (TTF) | from randomization to discontinuation of treatment for any reason, including progressive disease, treatment toxicity and death, assessed up to 48 months
  TTF will be defined as the time from randomization to discontinuation of treatment for any reason, including progressive disease, treatment toxicity and death; in the absence of treatment failure time will be censored at the last known follow-up.
Objective Response Rate (ORR) | up to 48 months
  ORR is defined as the percentage of patients achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria
Disease Control Rate (DCR) | Up to approximately 48 months
  DCR is defined as the percentage of patients achieving a complete (CR) or partial (PR) response or a stable disease (SD), according to RECIST 1.1 criteria
Quality of life (QoL) | Up to approximately 48 months
  QoL will be estimated with EORTC QLQ-C30 and the modules PAN26, FA12, CAX24, COMU26 a will be performed with the EORTC QLQ INFO25, which is a valid self-reported instrument consisting of 25 questions. Communication between patients and professionals will be assessed with the EORT QLC COMU26.
Toxicity rate | Up to approximately 48 months
  Toxicity is defined as the percentage of patients experiencing a specific adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0).
Proportion of patients not eligible to randomization | Up to approximately 48 months
  Proportion of patients not eligible to randomization is defined as patients who started induction treatment but result not eligible due to i) clinical deterioration or treatment toxicity, ii) withdraw consent or iii) disease progression documented as best response, iv) other causes
Subsequent treatment line frequency | Up to approximately 48 months
  Subsequent treatment line frequency is defined as the percentage of patients who undergo a systemic treatment (excluding locoregional treatments or surgical treatment of unresectable disease) after progression to first line in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Monica Niger, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (28):
- Italy (28):
  - Centro Di Riferimento Oncologico Di Aviano, Aviano, Italy
  - University Hospital Consorziale Policlinico, Bari, Italy
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia, Italy
  - ASST Ospedale Maggiore di Crema, Crema, Italy
  - Azienda Socio Sanitaria Territoriale Di Cremona, Cremona, Italy
  - Careggi University Hospital, Florence, Italy
  - IRCCS Ospedale Policlinico San Martino, Genoa, Italy
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST S.r.l., Meldola, Italy
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Italy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
  - Istituto Europeo Di Oncologia S.r.l., Milan, Italy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy
  - Humanitas Istituto Clinico Catanese S.p.A., Misterbianco, Italy
  - Azienda Sanitaria Locale Napoli 1 Centro, Napoli, Italy
  - Azienda Ospedaliero-Universitaria Maggiore Della Carità, Novara, Italy
  - Istituto Oncologico Veneto, Padua, Italy
  - Azienda Ospedaliero Universitaria Parma, Parma, Italy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
  - Azienda Sanitaria Territoriale Di Pesaro E Urbino, Pesaro, Italy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Italy
  - Azienda Sanitaria Locale Della Provincia Di Biella, Ponderano, Italy
  - Azienda USL Toscana Centro, Prato, Italy
  - Azienda Unita Sanitaria Locale Della Romagna, Ravenna, Italy
  - I.F.O. Istituti Fisioterapici Ospitalieri, Rome, Italy
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy
  - Humanitas Mirasole S.p.A., Rozzano, Italy
  - Pia Fondazione Di Culto E Religione Cardinale Giovanni Panico, Tricase, Italy
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sciortino C, Nichetti F, Bergamo F, Palermo F, Tamberi S, Vivaldi C, Ongaro E, Arcangeli G, Marchesi S, Giommoni E, Cella CA, Pircher C, Chiaramonte A, Bencardino K, Sottotetti E, Martinetti A, Rapposelli IG, Corallo S, Di Donato S, Murialdo R, Delliponti L, Salvatore L, Bozzarelli S, Dell'Aquila E, Miceli R, Carnaghi C, Tomasello G, Rivizzigno P, Bonomi M, Mannavola F, Forti L, Garajova I, Attademo L, Galassi B, Chiari R, Leone F, Garattini SK, Tamburini E, Pietrantonio F, Niger M. A phase III randomized clinical trial of Gemcitabine and Nab-Paclitaxel as switch maintenance versus continuation of modified FOLFIRINOX as first-line chemotherapy in patients with advanced pancreatic cancer: The PANThEON Study. Dig Liver Dis. 2025 Dec;57(12):2470-2477. doi: 10.1016/j.dld.2025.11.007. Epub 2025 Nov 28. PMID 41318310